CLINICAL TRIAL: NCT05031910
Title: Preoperative Virtual Reality and 3D Pathologic Modeling as Treatment for Head and Neck Squamous Cell Carcinoma
Brief Title: Virtual Reality 3D-Surgery Modeling to Enhance Head and Neck Cancer Surgery Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21D.079; JT 15475 (Other: JeffTrial Number)
Record Dates: First submitted 2021-08-31; First posted 2021-09-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (VR/3D-CEPs, standard treatment) (Experimental): Prior to surgery (day 0-13), patients undergo virtual reality 3D tumor resection via VR/3D-CEPs. Patients' pre-surgical CT scans are reviewed per standard of care. Patients then undergo surgical resection on day 14-29 and a 3D model of true tumor is created and imported into the virtual reality environment.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Best Practice; Procedure: Resection
- Arm II (standard treatment) (Active Comparator): Prior to surgery (day 0-13), patients' pre-surgical CT scans are reviewed per standard of care. Patients then undergo surgical resection on day 14-29.
  Interventions: Other: Best Practice; Procedure: Resection

INTERVENTIONS:
Other: Medical Device Usage and Evaluation — Undergo virtual reality imaging via VR/3D-CEPs
  Arms: Arm I (VR/3D-CEPs, standard treatment)
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection

SUMMARY:
This clinical trial studies the use of virtual reality technology and three dimensional surgery (3D-surgery) modeling to enhance current treatments in head and neck cancer surgery. Virtual reality 3D-surgery modeling may improve quality of surgical planning and interdisciplinary communication between surgeons and pathologists during the treatment of head and neck squamous cell cancer and ultimately increase the accuracy of planning, the quality of communication, and maximize the outcome patients with head and neck cancer experience throughout treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To assess the potential for preoperative virtual reality and 3D pathological modeling to reduce total number of margin events as defined in the study as the number of positive frozen margins, number of positive final margins and the number of unexpected defect driven margins.

SECONDARY OBJECTIVES:

To assess the impact of preoperative virtual reality and 3D pathologic modeling as treatment for head and neck squamous cell carcinoma on event free survival (EFS) at 18-36 months after resection as defined by recurrence at the primary site.

TERTIARY OBJECTIVE:

I. To evaluate the quality of existing interdisciplinary intraoperative communication using the proposed VR/3D-case enhancement protocols (CEPs) as an evaluating medium.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (VR/3D-CEPs + STANDARD TREATMENT): Prior to surgery (day 0-13), patients undergo virtual reality 3D tumor resection via VR/3D-CEPs. Patients' pre-surgical computed tomography (CT) scans are reviewed per standard of care. Patients then undergo surgical resection on day 14-29 and a 3D model of true tumor is created and imported into the virtual reality environment.

ARM II (STANDARD TREATMENT): Prior to surgery (day 0-13), patients' pre-surgical CT scans are reviewed per standard of care. Patients then undergo surgical resection on day 14-29.

After completion of study intervention, patients are followed for up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer of the head and neck (oral cavity, oropharynx, larynx, hypopharynx, T1-T4)
* Receiving treatment at Thomas Jefferson University - Center City by a fellowship-trained HNC surgeon
* Eligible for definitive resection
* Age > 18
* Provide signed written informed consent document

Exclusion Criteria:

* Impaired judgement or those unable to provide informed consent
* Any factor that would place the patient at increased risk or preclude the individual's full compliance with or completion of the study
* Nasopharyngeal carcinoma
* Contraindications for surgery
* Enrollment in other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Margin events | Up to Completion of surgical resection
  Will be defined as the number of positive margins along with the number of unexpected defect driven margins. Will be collected for patients in the control group and patients treated with the use of preoperative planning with virtual reality (VR). Margin events will be defined as binary (yes/no) on post-operative survey to be completed by surgeons. Logistic regression will be used to evaluate of a difference in any margin event between study groups (3 dimensional [3D] VR vs. control) adjusted for surgeon.

SECONDARY OUTCOMES:
Event free survival | The time from completion of treatment to marginal recurrence of tumor at the primary site, assessed up to 3 years
  Logistic regression will be used to estimate an odds ratio and 95% confidence interval (CI).

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No